CLINICAL TRIAL: NCT05587348
Title: PROmoting Diabetes Education and Management Through Peer Support and Team Referral
Acronym: PROMPT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 22-0357; R34DK132571-01 (NIH)
Record Dates: First submitted 2022-10-14; First posted 2022-10-20 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Diabetes Self Management Education and Support; Peer Support
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 1. Best Practice Advisory (Experimental): Four practices receive a suite of tools intended to increase the rate of referral to DSMES classes for patients with type 2 diabetes. In these four practices, the assigned DCE specialist will have access to a list of eligible patients who have upcoming appointments with their primary care providers. The DCE specialist will message the providers about the eligible patients via the EHR. They will also place a pended order for referral to DSMES class for the eligible patients. The health care provider will be able to either approve or deny the order for the referral Additionally, when an eligible patient presents for an appointment in one of the four intervention clinics, a best practice advisory (BPA) will fire within the EHR and encourage the provider to place a referral for DSMES classes.
  Interventions: Behavioral: Best Practice Advisory
- 2. Silent Best Practice Advisory (Placebo Comparator): Two practices will not receive the suite of tools, but the lists and BPA will be created and sent to the research team.
  Interventions: Behavioral: Best Practice Advisory
- 3. Peer Support (Experimental): 45 patients in the 6 clinics who are referred to DSMES classes who enroll in the study will be assigned a peer supporter who will work with the participant and encourage attendance to the DSMES classes in addition to the usual support offered by the clinic.
  Interventions: Behavioral: Peer Support
- 4. Usual Care (Placebo Comparator): 45 patients in the 6 clinics who are referred to DSMES classes who enroll in the study will receive the usual support offered by the clinic.
  Interventions: Behavioral: Peer Support

INTERVENTIONS:
Behavioral: Best Practice Advisory — Provider will get Best Practice Advisory or Message from DCE in intervention practices
  Arms: 1. Best Practice Advisory; 2. Silent Best Practice Advisory
Behavioral: Peer Support — Patients referred to DSMES classes will be randomized to get a peer supporter
  Arms: 3. Peer Support; 4. Usual Care

SUMMARY:
A 3-step project is proposed. Step 1 will test which BPA time point(s) maximize referral rates to DSMES services in the real world clinic setting (Aim 1). Step 2 will utilize that approach within a pilot study of six sites, comparing the effectiveness of peer support to improve attendance to DSMES services (Aim 2). Step 3 will engage stakeholders in designing a future large scale DSMES services trial to improve referral and attendance to DSMES classes.

DETAILED DESCRIPTION:
Living with diabetes can be challenging, however Diabetes Self-Management Education and Support (DSMES) is well known to help persons with diabetes (PWDM) learn to cope with the uncertainties of life with diabetes. Unfortunately, DSMES is underutilized in the current health care setting. This is a multifactorial problem with the two largest issues being providers not referring patients and patients not attending the DSMES programs. These programs and the health care workers who support them have the potential to modify the disease course for many PWDM, including potentially modifying long term morbidity and mortality. A feasibility study to test the impact of best practice advisories (BPAs) delivered to the health care provider and the diabetes care and education (DCE) specialists via the electronic health record when a PWDM is identified as qualifying for DSMES. The investigators will determine if the BPAs influence the time to referral for DSMES as well as the factors that predict whether a patient is referred to DSMES. The investigators also propose to assess the impact of a peer support on motivating PWDM to attend DSMES and make healthier lifestyle choices. The investigators hypothesize that if PWDM are able to connect with a peer who is also living with diabetes, they may be more likely to attend DSMES. Finally, the investigators will assess qualitatively how the health care providers felt about the use of the BPA reminders, explore how the PWDM felt about the utility of the peer supporters, and the overall relevance of the diabetes education they received. From these lessons learned the investigators will work with the stakeholders to design a large, pragmatic randomized trial designed to increase the uptake of DSMES, a vital piece of the diabetes puzzle.

Aim 1. Evaluate the relative impact of BPAs on DSMES services among providers at 6 primary care clinics.The investigators will identify six primary care practices to deploy the suite of tools designed to increase patient referrals to DSMES classes. All six practices will be from within the state of North Carolina. The providers will be a mix of genders, and ages. Providers will be a convenience sample based upon the six practices that are identified to be a part of this study.

Aim 2. Conduct a 6-month pilot of DSMES among 90 PWDM randomized to one of two groups: usual care or peer support. The investigators will identify 90 PWD who are active adult patients with type 2 diabetes from one of the six practices identified in Aim 1.

Aim 3. Engage stakeholders in designing a future large scale DSMES services trial. The investigators will interview providers and patients from Aims 1 and 2 for the qualitative interviews planned in Aim 3.

Practices: Six primary care practices within the UNC Physicians Network (UNCPN) will be recruited. Based upon the strong relationship the investigators have built with the UNCPN over the past decade, the investigators will work with the UNCPN leadership team to identify practices most likely to be interested in participation. The investigators will ensure a diverse group of practices, including a mix of rural and urban locations. Upon identification of the potential practices, the seasoned practice facilitator will arrange lunch and learn sessions within the potential practices, where they will present the project and discuss the requirements of participating. Practices will have the opportunity to discuss participation amongst their team members, and the practice facilitator will follow up with them within a week to determine their interest in enrolling.

Patients: Patients who have been referred for DSMES classes will be consented and randomized to peer support or usual care. PWDM who are randomized to the peer support group will have standard DSMES classes and as well as support via a peer supporter. The no peer support group will receive standard DSMES class only. After a referral for DSMES class has been placed, the research team will contact them to discuss the pilot trial. Multiple recruitment approaches will be used including phone call, letter, email contact via Epic, the EPIC patient portal (MyChart) and informational flyers. Patients will be compensated for filling out surveys at baseline, 3 months, 6 months, and for optional focus group participation..

ELIGIBILITY:
Inclusion Criteria Providers:

* Primary Care Providers employed at the participating practices

Exclusion Criteria Providers:

* Primary Care Providers that are not employed at the participating practices

Inclusion Criteria Patients:

* Adult, English-speaking patients diagnosed with type 2 diabetes who are referred to DSMES classes from a provider at one of the study practices.

Exclusion Criteria Patients:

* Any patients who are not referred to DSMES classes from the study practices

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2023-09-12 (Actual); Primary Completion 2025-07-14 (Actual); Study Completion 2025-10-14 (Actual)

PRIMARY OUTCOMES:
Odds of referral for DSMES Placed through the Electronic Health Record (EHR) | 30 days
  EHR data from the Carolina Data Warehouse. Referral defined as within 30 days of patient seen in of office
Odds of attending 1 DSMES class | 3 months
  EHR data -odds of attending 1 DSMES class within 3 months of referral

SECONDARY OUTCOMES:
Time from index patient visit to referral to DSMES | 3 months
  EHR data- number of days from patient visit to referral placed in EMR
Time to get to DSMES class | 3 months
  EHR data- number of days from patient visit to attending DSMES class
Number of PWD who attended at least 2 DSMES group classes | 3 months
  EHR data - patients who attended two DSMES classes
Number of PWD who completed the entire DSMES class | 3 months
  EHR data - patients who attended the entire DSMES class series
A1c - Baseline | Baseline
  Pulled from EHR data
Change in A1c from baseline to 3 months | Baseline, Month 3
  Pulled from EHR data
Change in A1c from baseline to 6 months | Baseline, Month 6
  Pulled from EHR data
Diabetes Distress - Baseline | Baseline
  The Diabetes Distress Scale (DDS17) is a 17-item questionnaire assessing the severity of problems of living with diabetes. Participants indicate the degree to which each item impacts their life on a 6-point scale where 1 = not a problem and 6 = a very serious problem. The scores are summed and divided by 17 to generate an average score that can range from 1 to 6. Scores of 3 or more are considered high distress.
  The DDS17 has 4 sub-scores.
  A. Emotional burden, uses items 1,4, 7, 10, and 14 summed and divided by 5 to generate an average score.
  B. Physician distress, uses items 2, 5, 11, and15 summed and divided by 4 to generate an average score.
  C. Regimen distress, uses item 6, 8, 3, 12, and 16 summed and divided by 5 to generate an average score.
  D. Interpersonal distress, uses item 9,13, and 17 summed and divided by 3 to generate an average score.
  .
Change in Diabetes Distress from baseline to 3 months | Baseline, Month 3
  The Diabetes Distress Scale (DDS17) is a 17-item questionnaire assessing the severity of problems of living with diabetes. Participants indicate the degree to which each item impacts their life on a 6-point scale where 1 = not a problem and 6 = a very serious problem. The scores are summed and divided by 17 to generate an average score that can range from 1 to 6. Scores of 3 or more are considered high distress.
  The DDS17 has 4 sub-scores.
  A. Emotional burden, uses items 1,4, 7, 10, and 14 summed and divided by 5 to generate an average score.
  B. Physician distress, uses items 2, 5, 11, and15 summed and divided by 4 to generate an average score.
  C. Regimen distress, uses item 6, 8, 3, 12, and 16 summed and divided by 5 to generate an average score.
  D. Interpersonal distress, uses item 9,13, and 17 summed and divided by 3 to generate an average score.
Change in Diabetes Distress from baseline to 6 months | Baseline, Month 6
  The Diabetes Distress Scale (DDS17) is a 17-item questionnaire assessing the severity of problems of living with diabetes. Participants indicate the degree to which each item impacts their life on a 6-point scale where 1 = not a problem and 6 = a very serious problem. The scores are summed and divided by 17 to generate an average score that can range from 1 to 6. Scores of 3 or more are considered high distress.
  The DDS17 has 4 sub-scores.
  A. Emotional burden, uses items 1,4, 7, 10, and 14 summed and divided by 5 to generate an average score.
  B. Physician distress, uses items 2, 5, 11, and15 summed and divided by 4 to generate an average score.
  C. Regimen distress, uses item 6, 8, 3, 12, and 16 summed and divided by 5 to generate an average score.
  D. Interpersonal distress, uses item 9,13, and 17 summed and divided by 3 to generate an average score.
Diabetes Self-Efficacy Baseline | Baseline
  The Diabetes Self-Efficacy Survey Short Form (DES-SF) is an 8-item questionnaire assessing the ability of a person to self-manage their diabetes. Participants indicate the degree to which they agree with each of the statements on a 5 point scale where 1 = strongly disagree and 5 = strongly agree. The scores are summed and divided by 8 to generate an average score that can range from 1 to 5, with 5 indicating increased self-efficacy.
Change in Diabetes Self-Efficacy from baseline to 3 months | Baseline, Month 3
  The Diabetes Self-Efficacy Survey Short Form (DES-SF) is an 8-item questionnaire assessing the ability of a person to self-manage their diabetes. Participants indicate the degree to which they agree with each of the statements on a 5 point scale where 1 = strongly disagree and 5 = strongly agree. The scores are summed and divided by 8 to generate an average score that can range from 1 to 5 with 5 indicating increased self-efficacy
Change in Diabetes Self-Efficacy from baseline to 6 months | Baseline, Month 6
  The Diabetes Self-Efficacy Survey Short Form (DES-SF) is an 8-item questionnaire assessing the ability of a person to self-manage their diabetes. Participants indicate the degree to which they agree with each of the statements on a 5 point scale where 1 = strongly disagree and 5 = strongly agree. The scores are summed and divided by 8 to generate an average score that can range from 1 to 5 with 5 indicating increased self-efficacy.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Young, MD, PhD, Principal Investigator — UNC Chapel Hill; Katrina Donahue, MD, MPH, Principal Investigator — UNC Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Deidentified individual data that supports the results will be shared beginning 9 and continuing for 36 months following publication.
Access Criteria: Investigator has approved IRB, IEC, or REB and an executed data use/sharing agreement with UNC.

DOCUMENTS (1):
  • Informed Consent Form (2022-06-01): https://cdn.clinicaltrials.gov/large-docs/48/NCT05587348/ICF_000.pdf